CLINICAL TRIAL: NCT03242772
Title: Impact of Combined Medication and Behavioral Treatment in Young Children With Comorbid ASD and ADHD
Brief Title: Impact of Combined Medication and Behavioral Treatment for ASD & ADHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study stopped recruitment of new participants due to COVID. A substudy was developed with adaptations to the main design.
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00085179; 1P50HD093074-01 (NIH)
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESDM informed parent coaching + Amphetamine (Active Comparator): Amphetamine regimen (11 weeks total duration) will begin 2 weeks prior to initiation of ESDM informed parent coaching (8 weekly sessions) and continue through the week 11 endpoint assessment. The drug is an orally dissolvable, extended-release form of d- and l-amphetamine.
  Interventions: Drug: Amphetamine; Behavioral: ESDM informed parent coaching
- ESDM informed parent coaching + Placebo Oral Tablet (Placebo Comparator): Placebo regimen (11 weeks total duration) will begin 2 weeks prior to initiation of ESDM informed parent coaching (8 weekly sessions) and continue through the week 11 endpoint assessment. The placebo contains no active drug and appears identical to the amphetamine (active drug).
  Interventions: Behavioral: ESDM informed parent coaching; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Amphetamine — Study drug will be administered in the morning. Treatment will be initiated at 1 tablet = 3.1 mg or 0 mg of mixed amphetamine. Doses will be flexibly titrated upward and may be decreased or stopped at any time.
  Other Names: Adzenys XR-ODT
  Arms: ESDM informed parent coaching + Amphetamine
Behavioral: ESDM informed parent coaching — All participants will receive 8 weekly parent child therapy sessions will be delivered by a therapist trained in parent coaching and ESDM principles and strategies and utilizing a therapy manual,(includes coaching for behavior management and handouts).
Drug: Placebo Oral Tablet — Matched placebo tablets will be administered in the morning and provided for 11 weeks . The tablets will be titrated in the same way as the active drug and may be stopped at any time.
  Arms: ESDM informed parent coaching + Placebo Oral Tablet

SUMMARY:
Children with comorbid autism spectrum disorder (ASD) and attention deficit hyperactivity disorder (ADHD) have significantly worse outcomes than those with either ASD alone or ADHD alone. Effective early treatments that account for ADHD symptoms have not been developed for young children with ASD+ADHD. The overarching goals of this randomized, placebo-controlled, phase 2, pilot study are to (1) evaluate a novel early intervention that pharmacologically addresses ADHD symptoms while providing an ASD-targeted behavioral intervention, and (2) identify changes in behavioral and neurophysiological activity that may underlie improved outcomes in children with comorbid ASD and ADHD ages 3-10 years. The primary aim of this study is to evaluate whether a stimulant treatment augments efficacy of an ASD specific form of parent child therapy based on the Early Start Denver Model called ESDM influenced Parent Coaching. Secondary aims are to determine the efficacy of combined intervention in improving ADHD symptoms and the efficacy, safety, and tolerability of Adzenys-XR-ODT in young children with ASD+ADHD. The study will also examine correlations between behavioral changes and state-of-the-art eye-gaze tracking (EGT) and electroencephalographic (EEG) biomarkers to elucidate key ways in which ADHD impacts attentional and neural functioning in ASD+ADHD, and to potentially identify new targets for intervention in children with ASD+ADHD. The study is about 8 months long and will involve screening, baseline assessment followed by 10- 11 weeks of study drug treatment (active or placebo) and 8 sessions of ESDM informed parent coaching beginning after 2 weeks of study drug treatment, primary endpoint assessments at ~11 weeks, AE follow-up by phone at ~week 13 and remote FU 24 weeks after baseline. Eligible participants will be randomly assigned to the active medication or placebo, Between weeks 11 to 24, it is expected that the parent will use the behavioral strategies they were coached in even though they will not receive parent coaching. Participants will be given the option to pursue ADHD medication outside of the research study after week 11 assessments.

DETAILED DESCRIPTION:
This randomized, placebo-controlled, Phase 2, single site, pilot study will evaluate the developmental impact of combined medication and behavioral treatment (COMB) versus placebo and behavioral treatment (BEH) in children with comorbid ASD +ADHD, who are between 36 and < 132 months of age. The active medication treatment will be an orally dissolvable, extended release amphetamine preparation (Adzenys-XR-ODT) administered from weeks 0-~11 and carefully titrated to the optimal dose using an algorithm that considers adverse events and improvement in attention symptoms with a flexible dose range of 1.55mg - 18.6mg/day. The target dose is 12.4mg/day. A placebo, matched to the active medication, will be titrated and adjusted using the same algorithm in the BEH arm. The provided behavioral treatment will be eight ~ hour long parent child therapy sessions of ESDM influenced parent coaching.

Approximately 48 participants will be randomly assigned to either the COMB or BEH treatment arms. To account for possible differences in attrition due to potential poor tolerability of Adzenys-XR-ODT, participants will be randomized in a 7 COMB to 6 BEH ratio. Treatment assignment will be provided by the Data Management and Analysis Core (DMAC)using computer generated algorithms.

The primary analyses will compare changes in outcomes between weeks 0 and 11 weeks. Exploratory analyses will explore changes between weeks 0 and 24.

The primary outcome measure is change in amount and quality of joint engagement between the child and the parent during a semi-structured, 6 minute parent child interaction task (PCIT), which reflects the core symptom domain targeted by P-ESDM: social communication.

Our key secondary outcomes will be changes in 1) the mean of the interview version of the VABS-3 socialization subscale and communication subscale standard scores and 2) clinician ratings of ADHD symptoms using the preschool ADHD-RS.

We will also assess the safety and tolerability of Adzenys-XR-ODT compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of a parent signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Aged 36 months to less than 132 months.
4. Diagnosed with both ASD and ADHD based consensus diagnosis informed by results of the Autism Diagnostic Observation Schedule 2nd edition (ADOS-2), Autism Diagnostic Interview - Revised (ADI-R), and a Standardized ADHD Diagnostic Interview and the MINI psychiatric diagnostic interview.
5. In good general health as evidenced by medical history and physical exam and review of safety labs and electrocardiogram.

Exclusion Criteria:

1. Recent use of prohibited psychoactive medication in close proximity of baseline assessments. See MOP for specific medications that are prohibited and washout procedures. Use of a monoamine oxidase inhibitor is prohibited within 14 days of baseline.
2. Known allergic reactions to amphetamines or components of Adzenys-XR-ODT.
3. Known history of sudden non-ischemic cardiac death in a first or second degree family member (sibling, parent, aunt, uncle, cousin or grandparent).
4. Personal history of significant cardiac abnormalities or disease, particularly rhythm abnormalities.
5. Significant visual, auditory or motor impairments that would preclude participation in ESDM-informed parent coaching or completion of key assessments.
6. Inability of the caregiver participating in P-ESDM and responding to questionnaires to fluently speak English.
7. Parent's participation in another parent coaching intervention on more than a monthly basis that may affect study provided therapy as determined by the PI or clinician.
8. Presence of any psychiatric conditions or psychiatric symptoms in addition to ASD and ADHD that would confound assessments and/or affect participation in the study as deemed by the PI or clinician.
9. Known genetic (e.g. Fragile X) or neurological syndrome or condition with established link to autism, but not events in which the link to ASD is less well known/established (e.g., 16p11.2 CNVs, CHD8 mutations, Trisomy 21, 22q deletion syndrome)
10. History of epilepsy or seizure disorder (except for history of simple febrile seizures or if the child is seizure free (regardless of seizure type) for the past year).
11. History of neonatal brain damage. (eg., with diagnoses hypoxic or ischemic event)
12. Any known environmental circumstances that is likely to account for the picture of autism in the proband (severe nutritional or psychological deprivation etc.)
13. Study clinician judgment that it is not in the best interests of the participant and/or the study for the child to participate.

Ages: 36 Months to 131 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2021-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Dawson, PhD, Principal Investigator — Duke; Linmarie Sikich, MD, Principal Investigator — Duke; Scott Kollins, PhD, Principal Investigator — Duke
Locations (1):
- Duke Center for Autism and Brain Development, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Through NDAR, core assessment and diagnostic data that is de-identified, including measures such as ADOS and Vineland.
Supporting Information: Study Protocol
Time Frame: 1 year after publication of the results for each of the specific aims or 3 years after the statistical analyses are completed
Access Criteria: determined by committee of researchers/administrator at NDAR
URL: https://nda.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred through our autism research registry, community events and Duke clinics
Pre-assignment Details: Confirmation of dual diagnosis was required prior to randomization
Period: Overall Study
Arm/Group | ESDM Informed Parent Coaching + Amphetamine | ESDM Informed Parent Coaching + Placebo Oral Tablet
Started | 9 | 9
Completed | 6 | 8
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESDM Informed Parent Coaching + Amphetamine | ESDM Informed Parent Coaching + Placebo Oral Tablet | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: months] | 86.83 (20.80) | 103.00 (18.88) | 94.92 (19.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 9 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 5 | 13
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Amount and Quality of Joint Engagement Between the Child and Parent During a Semi-structured 6 Minute Parent Child Interaction Task
Description: Child engagement states measured by the Joint Engagement Rating Inventory (JERI); our outcome contains four items (rated on a 7-point Likert scale) that characterize various aspects of engagement. Higher scores mean greater/higher quality engagement and lower scores represent less/poorer engagement. Total range of score is 4-28.
Time Frame: Baseline (Week -1), Endpoint (Week 10)
Population: This variable required behavioral coding of videotaped caregiver-child interactions collected at two time points. This coding were not conducted due to the fact that the study was terminated and time 2 data were not collected for participants due to safety concerns related to Covid-19.
Arm/Group | ESDM Informed Parent Coaching + Amphetamine | ESDM Informed Parent Coaching + Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Mean Composite Score (Socialization and Communication Subscales Standard Scores) of the Vineland Adaptive Behavior Scale - 3rd Edition, Interview Version (VABS-3)
Description: Mean of standard scores for VABS-3 (socialization subscale and communication subscales) assess how the participant actually has been functioning over the preceding month with regard to communication and social behaviors. The VABS-3 comprehensive form will be administered as a semi-structured interview by a trained and research reliable staff member. The standard score is based on the participant's age and is normed from a large sample of typically developing children. The standard score has a mean of 100 and a standard deviation of 15. The composite score range is 20-140; higher scores represent more adaptive functioning and lower scores represent less adaptive functioning.
Time Frame: Baseline (Week -1), Endpoint (Week 10)
Population: Not all participants completed all surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESDM Informed Parent Coaching + Amphetamine | ESDM Informed Parent Coaching + Placebo Oral Tablet
Number analyzed (Participants) | 6 | 7
score on a scale | 5.92 (5.34) | 1.86 (6.89)
Statistical Analysis 1: Comparison: ESDM Informed Parent Coaching + Amphetamine vs ESDM Informed Parent Coaching + Placebo Oral Tablet; Test type: Other; p = 0.2664, 95% confidence interval — Significance at <0.05; confidence interval (CI) = -3.5729 - 11.6929; Presentation of results will include p-values and 95% confidence intervals for the least mean square values at weeks 0, 10, 24 (week 24 is exploratory)

3. Secondary Outcome: Change in ADHD Symptoms Using Preschool or School Age ADHD Rating Scale (ADHD-RS) Total Score
Description: ADHD Rating Scale (ADHD-RS) will assess symptom frequency using data from clinician completed ADHD-RS and parent completed ADHD-RS. The ADHD-RS includes 18 items, each rated on a 4 point scale (0-3);Total Score is the sum of all responses (0-54). An Inattention subscale and Hyperactivity/Impulsivity subscale (each range 0-27) are calculated based on individual items assessing those symptoms. Higher values represent worse outcomes for the subscales and the total scale. Clinically significant scores in boys are 14 for inattention and 17 for hyperactivity/impulsivity items; thresholds in girls are 12 and 14 respectively. If subscales are used, they would be summed to compute the total score. *Baseline measures occur on visits weeks -1 and week 0 in the study.
Time Frame: Baseline (Week 0), Week 10
Population: Not all participants completed all surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESDM Informed Parent Coaching + Amphetamine | ESDM Informed Parent Coaching + Placebo Oral Tablet
Number analyzed (Participants) | 4 | 8
score on a scale | -10.00 (6.81) | -4.75 (10.02)
Statistical Analysis 1: Comparison: ESDM Informed Parent Coaching + Amphetamine vs ESDM Informed Parent Coaching + Placebo Oral Tablet; Test type: Other; p = 0.3721, 95% confidence interval — Significance at <0.05; confidence interval (CI) = -17.7698 - 7.2698; [other analysis details as in outcome 2, analysis 1]

4. Secondary Outcome: Changes in Objective Measures of Social Attention and Social Engagement Using Eye Gaze Tracking
Description: Eye Gaze Tracking (EGT) during presentation of social and nonsocial stimuli. Key measure used is Proportion Looking Time, which is a number between 0 and 1, with a higher number indicating improved attention.
Time Frame: Baseline (Week -1), Week 10
Population: This variable required processing of eye tracking data collected at two time points. We chose not to process the eye tracking data due to the fact that the study was terminated and time 2 data were not collected for participants because of safety concerns related to Covid-19.
Arm/Group | ESDM Informed Parent Coaching + Amphetamine | ESDM Informed Parent Coaching + Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: First three participants had a time frame of 52-64 weeks, and the remaining 15 had a timeframe 24 weeks, per protocol.
Description: First three participants were systematic using the SLAES, next 15 subjects were spontaneous (non-systematic).
Arm/Group | ESDM Informed Parent Coaching + Amphetamine | ESDM Informed Parent Coaching + Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 9/9 | 8/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ESDM Informed Parent Coaching + Amphetamine (N=9) | ESDM Informed Parent Coaching + Placebo Oral Tablet (N=9)
Mood Dysregulation (Psychiatric disorders) | 5 | 4 — Mood Dysregulation includes verbatim reports of mood changes, poor coping, and low frustration tolerance.
Insomnia (Psychiatric disorders) | 5 | 1
Aggression (Psychiatric disorders) | 2 | 1
Compulsions (Psychiatric disorders) | 2 | 0
Hyperfocused (Psychiatric disorders) | 1 | 0
Stereotypies, worsened (Psychiatric disorders) | 1 | 0
Hyperactivity, worsened (Psychiatric disorders) | 1 | 0
Flat affect, worsened (Psychiatric disorders) | 1 | 0
Oppositionality, worsened (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Subjective Temperature Dysregulation (Nervous system disorders) | 1 | 0
Decreased Appetite (General disorders) | 2 | 1
Viral Infections (Infections and infestations) | 4 | 7
Accidental Injury (Injury, poisoning and procedural complications) | 1 | 0
Environmental Allergies, worsened (Immune system disorders) | 3 | 0
Inflamed Toe (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Constipation, increased (Gastrointestinal disorders) | 1 | 1
Motion Sickness (Ear and labyrinth disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruitis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT03242772/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT03242772/ICF_001.pdf